CLINICAL TRIAL: NCT01538615
Title: Healthy Home Offerings Via the Mealtime Environment (HOME) Plus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20521; R01DK084000-01A2 (NIH)
Record Dates: First submitted 2012-01-17; First posted 2012-02-24 (Estimated); Results first posted 2018-03-01 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-01

CONDITIONS: Obesity
Keywords: Family meals; Home food environment; Electronic media
MeSH Terms: conditions — Obesity | interventions — Methods

STUDY DESIGN:
Masking Description: This is a behavioral intervention. Masking is not feasible.
Oversight: Data Monitoring Committee: No

ARMS (2):
- HOME Plus Intervention (Experimental): described below
  Interventions: Behavioral: HOME Plus intervention
- Control (No Intervention): Control participants receive a monthly newsletter for the 10 months of the study with tips on healthy eating. The topics do not overlap the intervention content.

INTERVENTIONS:
Behavioral: HOME Plus intervention — The HOME Plus program families will participate in monthly, two-hour group sessions for ten months at local community centers. Each session offers new ideas focusing on family meals, healthy eating, and reducing sedentary behavior. At each session, families prepare and eat a meal together and participate in small group discussions and activities for both parent and child groups to promote healthy behaviors in the home. Topics include planning healthy meals and snacks with your family, having meals with your family more often, and improving the healthfulness of the food available at home. Families also receive periodic supportive phone calls throughout the year using motivational interviewing techniques to promote healthy behaviors to prevent and reduce childhood obesity.
  Arms: HOME Plus Intervention

SUMMARY:
The goal of the proposed project is to see if an innovative family-based intervention can reduce childhood obesity by actively engaging the whole family in promoting healthy behaviors in the home. In additions, the project will also examine how the HOME Plus family intervention influences children's dietary intake, frequency of family meals, availability of healthy and unhealthy foods in the home and served at meals and snacks, and screen time (TV, game systems). The study will provide important information on strategies that families can use at home to prevent obesity.

DETAILED DESCRIPTION:
Childhood obesity is a serious public health problem with limited effective prevention strategies to date. Although previous nutrition and physical activity environmental approaches for obesity prevention show some promise, most studies have not shown reductions in excess weight gain. Moreover, few prevention studies significantly engage parents and focus on the home environment. To prevent childhood obesity it is essential to promote healthy behaviors in the home environment because parents are influential primary role models for healthy eating and sedentary behavior, and are gatekeepers for food and beverage availability and degree of inactivity within the home. Moreover, the home setting is where most of children's calories and energy dense foods are consumed and where children engage in much of their sedentary behavior, particularly screen time (e.g., television, computer, game system). The proposed study will test the efficacy of the Healthy Home Offerings via the Mealtime Environment (HOME) Plus program, a ten-month, family-based health promotion intervention to prevent excess weight gain among 8-12 year old children. The program is based on Social Cognitive Theory and a socio-ecological framework and promotes both regular and nutritionally-sound snacks and meals in which family members eat together (i.e., family meals) and encourages reductions in sedentary behavior, particularly screen time among children in the home setting. The efficacy of the intervention will be tested in a randomized controlled trial with 160 families randomized to two conditions (intervention or attention-only control). Two cohorts of families, recruited from after-school programs and community centers, will be followed for 2.5 years. The primary hypothesis is that, by the end of the ten month intervention, target children in the intervention families, relative to children in the control families, will have significantly lower body mass index (BMI; primary outcome) after adjustment for baseline BMI values. Secondary outcomes include frequency of weekly family meals and number of healthful foods and beverages available in the home and served at family meals and snacks (as reported by parent), target children's daily intakes of healthful foods and beverages, and target children's minutes of sedentary behavior per week, particularly screen time. Child and parent measurement will occur in their homes at baseline, post-intervention (12-months post-randomization), and follow-up (9-months post-intervention) by trained research staff. The proposed study builds upon successful methods from our HOME pilot study (2006-2008; NIH R21-DK0072997) and is innovative as it actively engages entire families in experiential activities and capitalizes on the home setting. The study will provide important information on environmental and behavioral strategies that families can use at home to prevent excess weight gain. The intervention program has high translation potential and is likely to be immediately useful to families of school-age children because it will be tested in real-world community settings and sustained across the state of Minnesota by the University of Minnesota's Extension Service.

ELIGIBILITY:
Inclusion Criteria:

* the target child is between the ages of 8-12 years
* the target adult parent or guardian is the primary food preparer in the home
* target child has an age and gender adjusted body mass index at or above the 50th percentile
* participants are willing to be randomized into one of two groups (intervention or control)
* target child must live with participating adult most of the time

Exclusion Criteria:

* participants plan to move out of the area in the next six months
* participants have a severe food allergy, limitation, or medical condition that prevents them from participating in the intervention
* participants do not speak and read in English

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2010-07; Primary Completion 2015-07 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jayne A Fulkerson, PhD, Principal Investigator — University of Minnesota, School of Nursing
Locations (1):
- University of Minnesota, School of Nursing, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fulkerson JA, Neumark-Sztainer D, Story M, Gurvich O, Kubik MY, Garwick A, Dudovitz B. The Healthy Home Offerings via the Mealtime Environment (HOME) Plus study: design and methods. Contemp Clin Trials. 2014 May;38(1):59-68. doi: 10.1016/j.cct.2014.01.006. Epub 2014 Jan 27. PMID 24480729
- [Result] Draxten M, Fulkerson JA, Friend S, Flattum CF, Schow R. Parental role modeling of fruits and vegetables at meals and snacks is associated with children's adequate consumption. Appetite. 2014 Jul;78:1-7. doi: 10.1016/j.appet.2014.02.017. Epub 2014 Mar 12. PMID 24630934
- [Result] Friend S, Fulkerson JA, Neumark-Sztainer D, Garwick A, Flattum CF, Draxten M. Comparing childhood meal frequency to current meal frequency, routines, and expectations among parents. J Fam Psychol. 2015 Feb;29(1):136-40. doi: 10.1037/fam0000046. Epub 2014 Dec 8. PMID 25485670
- [Result] Flattum C, Draxten M, Horning M, Fulkerson JA, Neumark-Sztainer D, Garwick A, Kubik MY, Story M. HOME Plus: Program design and implementation of a family-focused, community-based intervention to promote the frequency and healthfulness of family meals, reduce children's sedentary behavior, and prevent obesity. Int J Behav Nutr Phys Act. 2015 Apr 29;12:53. doi: 10.1186/s12966-015-0211-7. PMID 25925226
- [Result] Fulkerson JA, Friend S, Flattum C, Horning M, Draxten M, Neumark-Sztainer D, Gurvich O, Story M, Garwick A, Kubik MY. Promoting healthful family meals to prevent obesity: HOME Plus, a randomized controlled trial. Int J Behav Nutr Phys Act. 2015 Dec 15;12:154. doi: 10.1186/s12966-015-0320-3. PMID 26667110
- [Result] Horning ML, Fulkerson JA, Friend SE, Neumark-Sztainer D. Associations among Nine Family Dinner Frequency Measures and Child Weight, Dietary, and Psychosocial Outcomes. J Acad Nutr Diet. 2016 Jun;116(6):991-9. doi: 10.1016/j.jand.2015.12.018. Epub 2016 Feb 10. PMID 26875023
- [Result] Draxten M, Flattum C, Fulkerson J. An Example of How to Supplement Goal Setting to Promote Behavior Change for Families Using Motivational Interviewing. Health Commun. 2016 Oct;31(10):1276-83. doi: 10.1080/10410236.2015.1062975. Epub 2016 Mar 3. PMID 26940585
- [Result] Loth KA, Friend S, Horning ML, Neumark-Sztainer D, Fulkerson JA. Directive and non-directive food-related parenting practices: Associations between an expanded conceptualization of food-related parenting practices and child dietary intake and weight outcomes. Appetite. 2016 Dec 1;107:188-195. doi: 10.1016/j.appet.2016.07.036. Epub 2016 Jul 31. PMID 27486926
- [Result] Horning ML, Fulkerson JA, Friend SE, Story M. Reasons Parents Buy Prepackaged, Processed Meals: It Is More Complicated Than "I Don't Have Time". J Nutr Educ Behav. 2017 Jan;49(1):60-66.e1. doi: 10.1016/j.jneb.2016.08.012. Epub 2016 Oct 12. PMID 27743860
- [Result] Kubik MY, Gurvich OV, Fulkerson JA. Association Between Parent Television-Viewing Practices and Setting Rules to Limit the Television-Viewing Time of Their 8- to 12-Year-Old Children, Minnesota, 2011-2015. Prev Chronic Dis. 2017 Jan 19;14:E06. doi: 10.5888/pcd14.160235. PMID 28103183
- [Derived] Lee J, Helgeson E, Horning ML, Elgesma KM, Kubik MY, Fulkerson JA. Food Insecurity and Changes in Diet Quality and Body Mass Index z-Scores Among Elementary School Students. Child Obes. 2024 Oct;20(7):508-516. doi: 10.1089/chi.2023.0185. Epub 2024 Mar 28. PMID 38546529
- [Derived] Lee J, Kubik MY, Fulkerson JA, Kohli N, Garwick AE. The Identification of Family Social Environment Typologies Using Latent Class Analysis: Implications for Future Family-Focused Research. J Fam Nurs. 2020 Feb;26(1):26-37. doi: 10.1177/1074840719894016. Epub 2019 Dec 25. PMID 31874588
- [Derived] Lee J, Kubik MY, Fulkerson JA. Diet Quality and Fruit, Vegetable, and Sugar-Sweetened Beverage Consumption by Household Food Insecurity among 8- to 12-Year-Old Children during Summer Months. J Acad Nutr Diet. 2019 Oct;119(10):1695-1702. doi: 10.1016/j.jand.2019.03.004. Epub 2019 May 2. PMID 31056369
- [Derived] Arcan C, Friend S, Flattum CF, Story M, Fulkerson JA. Fill "half your child's plate with fruits and vegetables": Correlations with food-related practices and the home food environment. Appetite. 2019 Feb 1;133:77-82. doi: 10.1016/j.appet.2018.10.017. Epub 2018 Oct 17. PMID 30339784
- [Derived] Myers ML, Fulkerson JA, Friend SE, Horning ML, Flattum CF. Case study: Behavior changes in the family-focused obesity prevention HOME Plus program. Public Health Nurs. 2018 Jul;35(4):299-306. doi: 10.1111/phn.12403. Epub 2018 Apr 6. PMID 29624720

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total study enrollment was 413. Of those, 93 were enrolled in focus groups designed to help develop an disseminate the study. The remaining 320 took part in the HOME Plus study as described 81 parent/child dyads were randomized into the intervention condition and 79 parent/child dyads were randomized into the control condition).
Period: Overall Study
Arm/Group | HOME Plus Intervention | Control
Started | 162 | 158
Completed | 140 | 146
Not Completed | 22 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HOME Plus Intervention | Control | Total
Number analyzed (Participants) | 162 | 158 | 320
Age, Customized [Mean (Standard Deviation); unit: years]
  mean child age | 10.5 (1.4) | 10.1 (1.4) | 10.4 (1.4)
  mean parent age | 41.3 (8.0) | 41.3 (7.4) | 41.3 (7.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  gender: Male | 48 | 45 | 93
  gender: Female | 114 | 113 | 227
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 11 | 20
  Not Hispanic or Latino | 153 | 147 | 300
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 6 | 8
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 27 | 52
  White | 119 | 113 | 232
  More than one race | 13 | 11 | 24
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 162 | 158 | 320
child BMIz [Mean (Standard Deviation); unit: Z-score] — Population: This row reports on the the child BMIz scores. Parent BMI will be reported in the following row.
  Z-score
    number analyzed (Participants) | 81 | 79 | 160
    (all) | 0.95 (0.78) | 1.02 (0.73) | 0.99 (0.75)
parent BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: This row reports on the values for parent BMI. Child BMIz were reported in the previous row.
  kg/m^2
    number analyzed (Participants) | 81 | 79 | 160
    (all) | 27.64 (7.14) | 29.64 (7.68) | 28.63 (7.46)
receiving economic assistance [Count of Participants; unit: Participants] | 72 | 52 | 124

OUTCOME MEASURES:

1. Primary Outcome: Change in Child Body Mass Index (BMI Z-score)
Description: Trained study staff will measure parent and child height and weight and use this to calculate body mass index (BMI). BMI values were than standardized for age and gender using CDC guidelines to obtain BMI z-scores. Analyses controlled for child age and parent education at baseline.
Time Frame: Change from Baseline at 12 and 21 months
Population: Numbers reported are for the child in the parent/child dyad. At post-intervention (12 months after baseline), 74 intervention children and 75 control children were measured. At follow-up (21 months after baseline) 70 intervention children and 73 control children were measured.
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | HOME Plus Intervention | Control
Number analyzed (Participants) | 74 | 75
z-score
  Post Intervention (12 months after baseline) | 0.95 (0.04) | 0.99 (0.04)
  Follow-up (21 months after baseline): number analyzed (Participants) | 70 | 73
  Follow-up (21 months after baseline) | 0.94 (0.04) | 1.01 (0.04)

2. Secondary Outcome: Change in Target Children's Daily Intakes of Fruits and Vegetables
Description: A trained interviewer will complete three 24-hour dietary recalls at each data collection time point with the child. The three days will be averaged to get an estimate of usual intake. Analyses controlled for child age and parent education at baseline.
Time Frame: Change from Baseline at 12 and 21 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: average servings
Arm/Group | HOME Plus Intervention | Control
Number analyzed (Participants) | 74 | 75
average servings
  Post Intervention (12 months after baseline) | 2.7 (0.19) | 2.5 (0.18)
  Follow-up (21 months after baseline): number analyzed (Participants) | 70 | 73
  Follow-up (21 months after baseline) | 2.5 (0.19) | 2.6 (0.18)

3. Secondary Outcome: Change in Target Children's Hours of Screen Time (Television Viewing, Video and Computer Game Playing) Per Week
Description: Screen time will be measured with survey questions asking children how many hours per day they spend doing each sedentary activity (such as watching TV, using the computer, playing video games). Separate questions will be asked for week days and weekend days then the will be weighted to determine the hours of sedentary activity per week. Analyses controlled for child age and parent education at baseline.
Time Frame: Change from Baseline at 12 and 21 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: hours per week
Arm/Group | HOME Plus Intervention | Control
Number analyzed (Participants) | 74 | 75
hours per week
  Post Intervention (12 months after baseline) | 33.0 (3.06) | 33.0 (3.00)
  Follow-up (21 months after baseline): number analyzed (Participants) | 70 | 73
  Follow-up (21 months after baseline) | 34.4 (3.13) | 41.7 (3.03)

4. Secondary Outcome: Change in Number of Fruits and Vegetables Available in the Home
Description: The HOME Food Inventory assesses which foods families currently have in their home from a list of items. Analyses controlled for child age and parent education.
Time Frame: Change from Baseline at 12 and 21 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: number of fruits and vegetables
Arm/Group | HOME Plus Intervention | Control
Number analyzed (Participants) | 74 | 75
number of fruits and vegetables
  Post Intervention (12 months after baseline) | 22.5 (0.88) | 20.4 (0.86)
  Follow-up (21 months after baseline): number analyzed (Participants) | 70 | 73
  Follow-up (21 months after baseline) | 21.6 (0.89) | 21.9 (0.86)

ADVERSE EVENTS:
Time Frame: Adverse events were collected while the intervention was being delivered, over a 2 year period total or for 1 year for each participant.
Arm/Group | HOME Plus Intervention | Control
Serious Adverse Events (participants affected / at risk) | 0/162 | 0/158
Other Adverse Events (participants affected / at risk) | 0/162 | 0/158

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes